CLINICAL TRIAL: NCT03923803
Title: Diagnostic Values of C-reactive Protein and Procalcitonin in Predicting Bacterial Infection in Acute Exacerbations of Chronic Obstructive Pulmonary Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doha Ismail Moussa, Principal investigator, Assiut University
Other Study IDs: CRPPC
Record Dates: First submitted 2019-04-18; First posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic obstructive pulmonary disease: patients with acutely exacerbated Chronic obstructive pulmonary disease admitted in chest department Assiut university hospital ,30 patients who revealed sputum culture and inflammatory markers suggesting infection exacerbation will be followed up
  Interventions: Diagnostic Test: C- reactive protein; Diagnostic Test: Pro calcitonin

INTERVENTIONS:
Diagnostic Test: C- reactive protein — the measurement will be done by chemileumeniscence
Diagnostic Test: Pro calcitonin — the measurement will be done by chemileumeniscence

SUMMARY:
Chronic obstructive pulmonary disease is a serious disease . Exacerbations of Chronic obstructive pulmonary disease is an acute worsening condition of Chronic obstructive pulmonary disease, which always accompanied by clinical symptoms such as, shortness of breath and increased production of sputum. Respiratory infection (bacteria or viruses or mixed) is thought to be the main cause in most exacerbations.

ELIGIBILITY:
Inclusion Criteria:

- Patients admitted to the hospital

Exclusion Criteria:

* patients with malignancies
* patients with other systemic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acutely exacerbated chronic obstructive pulmonary disease
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
The level of C-reactive protein between Infection and Non-infectious inflammatory response in acute exacerbations of Chronic obstructive pulmonary disease patients | 24 hours
  Patients will be classified into cases with Infection or non-infectious inflammatory response according to the level of C-reactive protein